CLINICAL TRIAL: NCT03213587
Title: Apatinib in Treating Patients With Recurrent or Metastatic Nasopharyngeal Carcinoma (NPC) Who Had Failed Prior Platinum Based Chemotherapy
Brief Title: Apatinib in Treating Patients With Recurrent or Metastatic Nasopharyngeal Carcinoma (NPC)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Chen Xiaozhong, Director,Department of radiation oncology, Principal Investigator, Clinical Professor, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZJCH-2017-126
Record Dates: First submitted 2017-07-03; First posted 2017-07-11 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- apatinib (Experimental)
  Interventions: Drug: Apatinib

INTERVENTIONS:
Drug: Apatinib — 500 mg qd p.o. and it should be continued until disease progression or intolerable toxicity or patients withdrawal of consent

SUMMARY:
To evaluate the efficacy and safety of apatinib in treating patients with recurrent or metastatic nasopharyngeal carcinoma who failed prior platinum based chemotherapy

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologic confirmed recurrent and/or metastatic nasopharyngeal carcinoma( NPC )
2. Have failed for ≥1 lines of platinum based chemotherapy
3. At least one measurable lesion according to the RECIST 1.1
4. ≥ 18 and ≤ 65 years of age
5. ECOG performance scale 0-2
6. Life expectancy of more than 3 months
7. Adequate hepatic, renal and hematologic functions (hemoglobin ≥ 90g/L, platelets ≥ 100×10^9/L, neutrophils ≥ 1.5×10^9/L, serum transaminase < 2.5×the upper limit of normal(ULN), (If liver metastases, serum transaminase< 5×the ULN), creatinine clearance rate > 60ml/min.
8. Signed and dated informed consent.

Exclusion Criteria:

1. Prior therapy with tyrosine kinase -inhibitor agent targeting at VEGFR and PDGFR
2. Before or at the same time any, second malignancies except cured basal cell carcinoma of skin and carcinoma in-situ of uterine cervix
3. Any factors that influence the usage of oral administration
4. Known Spinal Cord compression or diseases of brain or pia mater by CT /MRI screening
5. Within 6 months before the first treatment occurs artery / venous thromboembolic events, such as cerebral vascular accident (including transient ischemic attack), deep vein thrombosis and pulmonary embolism, etc.
6. Within 3 months before the first treatment occurs myocardial infarction, unstable angina pectoris, cardiac angioplasty or stent implantation
7. Within 1 months before the first treatment received surgical operation and the wounds were not healed
8. Application of anticoagulants or vitamin K antagonists such as warfarin, heparin or its analogues; If the prothrombin time international normalized ratio (INR) ≤ 1.5, with the purpose of prevention, the use of small doses of warfarin (1mg orally, once daily) or low-dose aspirin (between 80mg to 100mg daily) is allowed
9. Blood coagulation abnormal, having hemorrhagic tendency (eg. active peptic ulcer disease) or receiving the therapy of thrombolysis or anticoagulation.
10. Preexisting serious accompanying disease which may bring great risk or influence the patient's compliance( uncontrolled hypertension, grade III - IV cardiac insufficiency, severe arrhythmia -QTc duration between 500 m/s, severe liver and kidney insufficiency :urine protein+ +, 24 hours urinary protein > 1.0 g, mental illness.)
11. history of organ transplants
12. Evidence of significant medical illness that in the investigator's judgment will substantially increase the risk associated with the subject's participation in and completion of the study.

    -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
CBR(Clinical Benefit Rate) | 12 weeks
  The sum rate of complete response, partial response and stable disease
The incidence of Grade 3-4 adverse events | 2 years
  Number of participants with adverse events and serious adverse events.In addition,estimating their relationship with apatinib.

SECONDARY OUTCOMES:
PFS (progression free survival) | 2 years
  from the first day of therapy to the date of disease progression or death from any cause, whichever was first (according the criterion of RECIST 1.1 ).
OS (overall survival) | 2 years
  from the first day of therapy to death or last follow-up
QoL(quality of life) | 2 years
  Changes in quality of life were assessed by EORTC QLQ-C30

CONTACTS AND LOCATIONS:
Locations (1):
- Xiaozhong Chen, Hangzhou, Zhejiang, China